Prolonged Daily Fasting As a Viable Alternative to Caloric Restriction in At-Risk Obese Humans

NCT04259632 **6/20/22** 

## STATISTICAL ANALYSIS

The primary hypothesis was that the TRE and CR groups would have similar weight loss relative to baseline, which would be greater than weight loss achieved in the UE group. The study was powered to detect differences in weight loss (randomization to 12 weeks) for TRE and CR relative to UE, while preserving type-1 error for pairwise comparisons across all three groups. Based on the preliminary data and the literature <sup>35</sup> we anticipated weight loss of 3.6 kg (1.9) [mean (SD)] with TRE, 4 kg (2.5) with CR, and 1.5 kg (2.4) with UE. With n=24 per group and alpha = 0.05/3 to adjust for multiple comparisons, we estimated 80% power to detect the described difference in weight loss between TRE vs UE and 85% power to detect the described difference in weight loss between CR group vs UE.

Data were analyzed by intention-to-treat. Pre-post intervention change in outcomes were compared between the three groups using linear regression models with pairwise comparisons conducted using Tukey's method to account for multiple comparisons. The primary efficacy analysis included all randomized individuals with missing outcome measures imputed using multivariate imputation by chained equations. As a sensitivity analysis, the primary outcome analysis was conducted using only individuals who had complete data for the outcome of interest. (Supplementary Table 1). An additional sensitivity analysis among study completers was conducted excluding one participant in the UE group who reported noncompliance and had extreme weight loss (14.1 kg).

Multivariate imputation by chained equations was conducted using predictive mean matching to impute the primary and secondary outcome variables (weight, whole body percent fat, visceral fat, lean mass, fat mass, calorie intake; M-Value from clamp low dose infusion, M-Value from clamp high dose infusion, metabolic flexibility at end of low-dose clamp, metabolic flexibility at end of high-dose clamp and resting energy expenditure. Auxiliary variables included in the imputation included study arm, days from randomization to body composition and clamp assessments, age, sex, and baseline systolic and diastolic blood pressure, fasting: LDL, HDL, triglycerides glucose, insulin, hemoglobin A1C, eating window and healthy eating index.

For the imputation of cardiometabolic measures (resting energy expenditure, HDL, triglycerides, LDL, HbA1c, HOMA-IR, fasting glucose, fasting insulin, and CGM measures) auxiliary variables included in the imputation

were study arm, days from randomization to study assessments, sex, age, baseline systolic and diastolic blood

pressure, and baseline weight. For the imputation of dietary and lifestyle measures (calories, HEI, servings of sugar sweetened beverages, and actigraphy measures of activity and sleep) auxiliary variables included study arm, days from randomization to study assessments, sex, age, baseline systolic and diastolic blood pressure, and baseline weight, eating window, fasting glucose, fasting insulin, HDL, triglycerides, and LDL, Linear model results for change in outcome were pooled across 50 imputations using Rubin's rules <sup>36</sup> for computing the total variance.

For representing change in measures using forest plots, outcomes were transformed into z-scores by subtracting the overall mean and dividing by the overall standard deviation prior to fitting the unadjusted linear regression model.

The association between change in eating window and pre-post intervention change in outcome among study completers in the TRE and UE groups was assessed using linear regression models. Eating window calculated using time frame encompassing 95% of eating occasions and change in eating window was calculated as difference in eating window from baseline (prior to randomization) and end-of-intervention (Weeks 10-12). The CR arm was not included in these analyses since they were not instructed to document all eating occasions for the duration of the study using the mCC app.

All analyses were carried out using R (Version 4.3.1, R Foundation for Statistical Computing, Vienna, Austria) or SAS (Version 9.4, SAS Institute Inc., Cary, NC).

## **REFERENCES:**

- Gill, S. & Panda, S. A Smartphone App Reveals Erratic Diurnal Eating Patterns in Humans that Can Be Modulated for Health Benefits. *Cell Metabolism* **22**, 789-798 (2015). https://doi.org/10.1016/j.cmet.2015.09.005
- Maguen, S. et al. Screen for Disordered Eating: Improving the accuracy of eating disorder screening in primary care. General Hospital Psychiatry 50, 20-25 (2018). https://doi.org/https://doi.org/10.1016/j.genhosppsych.2017.09.004
- Leech, R. M., Worsley, A., Timperio, A. & McNaughton, S. A. Characterizing eating patterns: a comparison of eating occasion definitions. *The American journal of clinical nutrition* **102**, 1229-1237 (2015). https://doi.org/10.3945/ajcn.115.114660
- Frankenfield, D., Roth-Yousey, L. & Compher, C. Comparison of predictive equations for resting metabolic rate in healthy nonobese and obese adults: a systematic review. *J Am Diet Assoc* **105**, 775-789 (2005). <a href="https://doi.org/10.1016/j.jada.2005.02.005">https://doi.org/10.1016/j.jada.2005.02.005</a>
- Association, A. o. N. a. D. a. t. A. D. *Choose Your Foods: Food Lists for Weight Management*. (Academy of Nutrition and Dietetics and the American Diabetes Association, 2019).
- 6 Kaul, S. *et al.* Dual-Energy X-Ray Absorptiometry for Quantification of Visceral Fat. *Obesity* **20**, 1313-1318 (2012). https://doi.org/10.1038/oby.2011.393
- Bosch, T. A. *et al.* Identification of Sex-Specific Thresholds for Accumulation of Visceral Adipose Tissue in Adults. *Obesity* **23**, 375-382 (2015). <a href="https://doi.org/10.1002/oby.20961">https://doi.org/10.1002/oby.20961</a>
- Yushkevich, P. A. *et al.* User-guided 3D active contour segmentation of anatomical structures: significantly improved efficiency and reliability. *Neuroimage* **31**, 1116-1128 (2006). https://doi.org/10.1016/j.neuroimage.2006.01.015
- Demerath, E. W. *et al.* Approximation of total visceral adipose tissue with a single magnetic resonance image. *The American journal of clinical nutrition* **85**, 362-368 (2007). https://doi.org/10.1093/ajcn/85.2.362
- Maislin, G. *et al.* Single slice vs. volumetric MR assessment of visceral adipose tissue: reliability and validity among the overweight and obese. *Obesity (Silver Spring, Md.)* **20**, 2124-2132 (2012). <a href="https://doi.org/10.1038/oby.2012.53">https://doi.org/10.1038/oby.2012.53</a>
- Malin, S. K. *et al.* Insulin sensitivity and metabolic flexibility following exercise training among different obese insulin-resistant phenotypes. *American Journal of Physiology-Endocrinology and Metabolism* **305**, E1292-E1298 (2013). https://doi.org/10.1152/ajpendo.00441.2013
- Friedewald, W. T., Levy, R. I. & Fredrickson, D. S. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. *Clin Chem* **18**, 499-502 (1972).
- Bonora, E. *et al.* Homeostasis model assessment closely mirrors the glucose clamp technique in the assessment of insulin sensitivity Studies in subjects with various degrees of glucose tolerance and insulin sensitivity. *Diabetes Care* **23**, 57-63 (2000).
- Bergenstal, R. M. et al. Recommendations for standardizing glucose reporting and analysis to optimize clinical decision making in diabetes: the ambulatory glucose profile. Journal of diabetes science and technology 7, 562-578 (2013). https://doi.org/10.1177/193229681300700234
- Migueles, J., Rowlands, A., Huber, F., Sabia, S. & van Hees, V. GGIR: A Research Community–Driven Open Source R Package for Generating Physical Activity and Sleep Outcomes From Multi-Day Raw Accelerometer Data. *Journal for the Measurement of Physical Behaviour* **2**, 188-196 (2019). https://doi.org/10.1123/jmpb.2018-0063
- van Hees, V. T. *et al.* Separating movement and gravity components in an acceleration signal and implications for the assessment of human daily physical activity. *PLoS One* **8**, e61691 (2013). <a href="https://doi.org/10.1371/journal.pone.0061691">https://doi.org/10.1371/journal.pone.0061691</a>

- Sabia, S. *et al.* Association between questionnaire- and accelerometer-assessed physical activity: the role of sociodemographic factors. *Am J Epidemiol* **179**, 781-790 (2014). https://doi.org/10.1093/aje/kwt330
- van Hees, V. T. *et al.* Estimating sleep parameters using an accelerometer without sleep diary. *Sci Rep* **8**, 12975 (2018). <a href="https://doi.org/10.1038/s41598-018-31266-z">https://doi.org/10.1038/s41598-018-31266-z</a>
- Hildebrand, M., VT, V. A. N. H., Hansen, B. H. & Ekelund, U. Age group comparability of raw accelerometer output from wrist- and hip-worn monitors. *Med. Sci. Sports Exerc.* **46**, 1816-1824 (2014). https://doi.org/10.1249/mss.00000000000000289
- Matthews, C. E. *et al.* Accelerometer-measured dose-response for physical activity, sedentary time, and mortality in US adults. *The American journal of clinical nutrition* **104**, 1424-1432 (2016). https://doi.org/10.3945/ajcn.116.135129
- Trost, S. G., Loprinzi, P. D., Moore, R. & Pfeiffer, K. A. Comparison of Accelerometer Cut Points for Predicting Activity Intensity in Youth. *Medicine and Science in Sports and Exercise* **43**, 1360-1368 (2011). https://doi.org/10.1249/MSS.0b013e318206476e
- Healy, G. N., Matthews, C. E., Dunstan, D. W., Winkler, E. A. H. & Owen, N. Sedentary time and cardio-metabolic biomarkers in US adults: NHANES 2003-06. *Eur. Heart J.* **32**, 590-597 (2011). <a href="https://doi.org/10.1093/eurheartj/ehq451">https://doi.org/10.1093/eurheartj/ehq451</a>
- Tucker, J. M., Welk, G. J. & Beyler, N. K. Physical Activity in US Adults Compliance with the Physical Activity Guidelines for Americans. *American Journal of Preventive Medicine* **40**, 454-461 (2011). <a href="https://doi.org/10.1016/j.amepre.2010.12.016">https://doi.org/10.1016/j.amepre.2010.12.016</a>
- Sadeh, A., Sharkey, K. M. & Carskadon, M. A. Activity-based sleep-wake identification: an empirical test of methodological issues. *Sleep* **17**, 201-207 (1994). https://doi.org/10.1093/sleep/17.3.201
- Sadeh, A., Hauri, P. J., Kripke, D. F. & Lavie, P. The role of actigraphy in the evaluation of sleep disorders. *Sleep* **18**, 288-302 (1995). https://doi.org/10.1093/sleep/18.4.288
- Cole, R. J., Kripke, D. F., Gruen, W., Mullaney, D. J. & Gillin, J. C. Automatic sleep/wake identification from wrist activity. *Sleep* 15, 461-469 (1992). https://doi.org/10.1093/sleep/15.5.461
- 27 Center, U. o. M. N. C. *Nutrition Data System for Research.*, (University of Minnesota Nutrition Coordinating Center).
- 28 Reedy, J. *et al.* Evaluation of the Healthy Eating Index-2015. *J Acad Nutr Diet* **118**, 1622-1633 (2018). https://doi.org/10.1016/j.jand.2018.05.019
- 29 Krebs-Smith, S. M. *et al.* Update of the Healthy Eating Index: HEI-2015. *J Acad Nutr Diet* **118**, 1591-1602 (2018). <a href="https://doi.org/10.1016/j.jand.2018.05.021">https://doi.org/10.1016/j.jand.2018.05.021</a>
- 30 Willett, W. & Willett, W. in *Nutritional Epidemiology* 0 (Oxford University Press, 2012).
- Flint, A., Raben, A., Blundell, J. E. & Astrup, A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. *Int J Obes Relat Metab Disord* **24**, 38-48 (2000). <a href="https://doi.org/10.1038/sj.ijo.0801083">https://doi.org/10.1038/sj.ijo.0801083</a>
- 32 Crose, A. *et al.* Time-Restricted Eating Improves Quality of Life Measures in Overweight Humans. *Nutrients* **13**, 1430 (2021).
- Ware, J. E., Kosinski, M. & Keller, S. D. A 12-item short-form health survey Construction of scales and preliminary tests of reliability and validity. *Medical Care* **34**, 220-233 (1996). https://doi.org/10.1097/00005650-199603000-00003
- Ware, J. E., Jr. SF-36 health survey update. *Spine (Phila Pa 1976)* **25**, 3130-3139 (2000). https://doi.org/10.1097/00007632-200012150-00008
- Chow, L. S. *et al.* Time-Restricted Eating Effects on Body Composition and Metabolic Measures in Humans who are Overweight: A Feasibility Study. *Obesity (Silver Spring, Md.)* **28**, 860-869 (2020). https://doi.org/10.1002/oby.22756
- Rubin, D. B. Multiple Imputation for Nonresponse in Surveys. (John Wiley & Sons, Inc., 1987).